CLINICAL TRIAL: NCT04247620
Title: DiaBetter Together: A Strengths-based, Peer Mentor Transition RCT for Young Adults With Type 1 Diabetes
Brief Title: DiaBetter Together for Young Adults With Type 1 Diabetes
Acronym: DiaBetter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Marisa Hilliard, Associate Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-45360; 1R01DK119246 (NIH)
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Peer Support; Adherence; Young Adult; Quality of Life; Transition; Resilience; Strengths-based; Sleep; COVID-19 Experiences
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: A parallel two-group design will be used to evaluate the intervention among n=150 young adults randomly assigned to the peer support intervention or usual care (1:1). All young adults are randomized to either an intervention group, in which they all receive the same treatment in addition to usual diabetes care, or a control group, in which they receive usual diabetes care without the additional intervention. Young adult participants will be in the study for 12 months.
  Peer Mentor participants (up to n=36) will deliver the intervention to young adults randomized to the intervention group, and their outcomes related to being a Peer Mentor will also be evaluated pre-post.
Who Masked: Outcomes Assessor
Masking Description: Participants will be aware of their assignment to intervention or control, as will the investigators. However, the person collecting HbA1c (primary outcome) at baseline and follow-up (12 mo) will not be aware of the participant's assignment in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DiaBetter Together Intervention (Experimental): Young Adult participants with type 1 diabetes (ages 17-25) who are approaching transfer from pediatric to adult care will be randomized to either the DiaBetter Together Intervention group or the Usual Care group. After randomization to the intervention group, young adults will be assigned a Peer Mentor. Following an intervention manual, the Peer Mentor will teach behavioral strategies and offer support to the young adult. In both conditions, participation in this study will not impact participants' ability to contact the pediatric TCH diabetes care team or any other medical services to receive medical care.
  Interventions: Behavioral: DiaBetter Together
- Peer Mentors (Other): Peer Mentors will deliver the DiaBetter Together intervention and will also be enrolled as study participants to permit assessment of their own outcomes from delivering this peer support intervention to younger people with diabetes. Peer Mentors will be experienced young adults with T1D who have transferred to adult diabetes care.
  Interventions: Behavioral: Peer Mentor Delivery
- Usual Care (No Intervention): Participants randomized to the comparison condition will receive usual diabetes care only, without additional intervention through the study. They will participate in all study activities related to data collection, but will not receive the Peer Mentor intervention. In both conditions, participation in this study will not impact participants' ability to contact the pediatric TCH diabetes care team or any other medical services to receive medical care.
- Research Supplement (No Intervention): Following completion of 12-month data collection, a subset of participants from the Usual Care group will have the opportunity to complete an optional and additional week (7 days) of follow-up data collection to characterize general and diabetes-specific sleep patterns.

INTERVENTIONS:
Behavioral: DiaBetter Together — Following an intervention manual, the Peer Mentor will teach behavioral strategies and offer support to the young adult, including (a) teaching and modeling strengths-based skills for goal-setting, problem-solving, and stress management; (b) guiding participants in obtaining support from their social support network (e.g., family, friends); (c) developing a plan for accountability around diabetes management and follow-up in adult care; (d) sharing his/her transition experiences and strategies for successfully navigating the adult healthcare system; (e) discussing how to prioritize diabetes self-care; and (f) assisting them in accessing diabetes-related resources (e.g., local diabetes groups, apps, social media). Contact will be in-person, by phone, email, text message, and/or video, approximately weekly for first 3 mos, approximately biweekly for next 3 mos, and approximately monthly for last 6 mos (while COVID-19 safety recommendations are in place, in-person meetings will not occur).
  Arms: DiaBetter Together Intervention
Behavioral: Peer Mentor Delivery — Peer Mentors deliver the intervention to multiple young adult participants, each for 12 months. Peer Mentors may take on one or more participants at a time, and Peer Mentors may stay in their role in the study (delivering the intervention) for 1-3 years.
  Arms: Peer Mentors

SUMMARY:
DiaBetter Together is a strengths-based peer support intervention delivered to young adults (age 17-25) by trained Peer Mentors (age 20-35) during the transition between pediatric and adult diabetes care. The aims of this proposed randomized controlled trial are to evaluate the impact of the intervention on glycemic control (primary), time to first adult care visit, adherence, and psychosocial outcomes (secondary) in young adults with T1D after 12 months.

DETAILED DESCRIPTION:
DiaBetter Together is a strengths based peer support intervention delivered to young adults (age 17-25) by trained Peer Mentors (age 20-35) during the transition between pediatric and adult diabetes care. The study aims to optimize transition in T1D by leveraging and building on young adults' diabetes strengths, self-management skills, and social supports. This intervention will maximize protective processes that can facilitate optimal transition by training Peer Mentors (experienced young adults with T1D who have successfully established care in an adult setting) to provide relevant information about successful transition, teach strengths-based skills for managing transition-related challenges, share personal transition-related experiences, encourage young adults to access their social support network, and serve as a positive role model. Delivery of these strengths-based intervention components through a Peer Mentor has potential to reduce isolation, increase access to relevant information, and facilitate engagement with self-management and T1D care. This intervention is a complement to existing systems of care for young adults with T1D for 12 months as they leave the pediatric setting.

ELIGIBILITY:
Young Adult Inclusion/Exclusion Criteria

Inclusion Criteria:

* has a diagnosis of type 1 diabetes of at least 1 year
* currently receiving care at a Texas Children's Hospital Diabetes Care Center location
* is between the ages of 17-25 years at enrollment
* exhibits fluency in reading/speaking English
* their endocrine provider confirmed plans to transfer to adult provider in the next 6 months

Exclusion Criteria:

* serious medical, cognitive, or mental health comorbidity that would preclude ability to provide informed consent or participate in data collection or intervention

Peer Mentor Inclusion/Exclusion Criteria

Inclusion Criteria:

* was diagnosed with type 1 diabetes before age 18
* has a diagnosis of type 1 diabetes of at least 1 years
* is between the ages of 20-35 at enrollment
* has been previously treated in pediatric care and is currently treated in adult care
* demonstrated interest and ability to effectively deliver the peer intervention &
* exhibits fluency in reading/speaking English

Exclusion Criteria:

* serious medical, cognitive, or mental health comorbidity that would preclude ability to fulfill role or complete questionnaires.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa E Hilliard, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants receive informed consent form, and other participant data is not returned to participant.
Supporting Information: ICF
Time Frame: Receive copy of signed informed consent form upon signing
Access Criteria: All participants receive copy of signed informed consent form

REFERENCES:
- [Derived] Macke CA, Carreon SA, Desai KR, Minard CG, Lyons SK, McKay S, Devaraj S, Streisand R, Tang T, Anderson BJ, Hilliard ME. COVID-19 vaccine uptake and attitudes in emerging adults with type 1 diabetes. Vaccine. 2025 Aug 13;61:127083. doi: 10.1016/j.vaccine.2025.127083. Epub 2025 Jul 31. PMID 40750525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 115 young adults consented to the trial. Of those, 14 did not complete baseline data and were therefore not randomized, and 1 was withdrawn due to a change in eligibility.
  29 peer mentors consented to the trial and completed baseline data.
Pre-assignment Details: Results reflect the number of participants who completed data. This differs from the protocol enrollment number, as some consented participants did not complete baseline data and thus were not randomized or followed for subsequent data collection.
  Following trial completion, a subset of 20 participants from the Usual Care group completed an additional week of data collection related to their experiences with sleep. No intervention was administered - data collection only.
Period: Overall Study
Arm/Group | DiaBetter Together Intervention | Usual Care | Peer Mentors
Started | 50 | 50 | 29
Sleep Supplement Participation | 0 | 20 | 0
Completed | 44 | 48 | 29
Not Completed | 6 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All Research Supplement participants were previously enrolled in trial, either DiaBetter Together or Usual Care arm
Groups:
- Total: Total of all reporting groups
Arm/Group | DiaBetter Together Intervention | Usual Care | Peer Mentors | Total
Number analyzed (Participants) | 50 | 50 | 29 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.0 (1.3) | 19.9 (1.3) | 25.1 (3.3) | 21.1 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 21 | 79
  Male | 17 | 25 | 8 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: African American/Black, non-Hispanic | 8 | 4 | 1 | 13
  Race and Ethnicity: American Indian/Alaska Native, non-Hispanic | 1 | 0 | 0 | 1
  Race and Ethnicity: Asian, non-Hispanic | 1 | 2 | 2 | 5
  Race and Ethnicity: Hispanic | 8 | 17 | 6 | 31
  Race and Ethnicity: White, non-Hispanic | 29 | 25 | 20 | 74
  Race and Ethnicity: Another or multiple | 3 | 2 | 0 | 5
Insurance [Count of Participants; unit: Participants] — Population: Self-reported health insurance type
  Participants
    Private or Commercial | 27 | 26 | 27 | 80
    Public, County, Other, or No Insurance | 18 | 16 | 2 | 36
    Unsure | 5 | 8 | 0 | 13
Insulin delivery method, self-reported [Count of Participants; unit: Participants]
  Insulin Pump | 27 | 29 | 25 | 81
  Injections | 23 | 21 | 4 | 48
Continuous glucose monitor use, self-reported [Count of Participants; unit: Participants] | 42 | 34 | 27 | 103

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control (HbA1c)
Description: HbA1c is the average blood glucose over 3-4 months. The American Diabetes Association recommends an HbA1c target of <7.0%. HbA1c is collected via fingerstick/blood assay at routine diabetes visits and will be extracted from the medical record at each clinic visit during the study period.
  At Baseline and 12 months, HbA1c will be collected using the following methods:
  1. Collection of most recent HbA1c from review of electronic medical chart (Texas Children's or Baylor College of Medicine) or medical records from outside provider (obtained with written permission from participant).
  2. A dried blood spot at-home Hemoglobin A1c kit (Whatman 903 card, BD Microtainer HI-Flow Contact-Activated Lancet) will be mailed to the participant to complete and return to the study team for analysis on the Vitros 4600 HbA1c assay (correlated with the DCA 2000).
  Collected for young adult participants in both arms. Peer mentors self-reported HbA1c at baseline only.
Time Frame: Baseline through 12-Month Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | DiaBetter Together Intervention | Peer Mentors | Usual Care
Number analyzed (Participants) | 50 | 29 | 50
Percentage of HbA1c
  Baseline | 9.1 (2.0) | 6.5 (0.7) | 8.5 (2.0)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 41 | 0 | 43
  End of Study at 12 Months Post-Randomization | 9.2 (2.3) |  | 8.6 (1.9)

2. Secondary Outcome: Time to First Adult Care Visit
Description: Time will start on the date of the last pediatric care visit (may differ from date of enrollment in study). The event of interest is the date of the first adult care visit. Participants who do not follow-up with an adult care provider within 12 months of the last pediatric visit will be censored for the event at the 12-month time point.
  Collected for young adult participants in both arms, not Peer Mentors.
Time Frame: End of Study at 12 Months Post-Randomization
Population: Time to adult care visit was unable to be collected for most trial participants
Measure: Mean (Standard Deviation); unit: month
Arm/Group | DiaBetter Together Intervention | Usual Care
Number analyzed (Participants) | 8 | 4
month | 4.7 (2.1) | 7.7 (2.9)

3. Secondary Outcome: Diabetes Self-Management/Adherence (Self-Care Inventory-Updated)
Description: The Self-Care Inventory-Updated (SCI-U) is a 8-item measure that asks respondents the frequency with which they completed diabetes self-management tasks in the past 1-2 months. Item responses range from (1) Never to (5) Always, higher scores = higher adherence. A total score is calculated by summing and averaging all items, with no subscales. The minimum possible score is 8 and the maximum possible score is 40. Higher scores indicate higher engagement in diabetes self-management behaviors.
  Collected for young adult participants in both arms (baseline, 6 mo, 12 mo) and Peer Mentors (pre- and post-involvement in study).
Time Frame: Baseline, 6-Month Post-Randomization, & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care | Peer Mentors
Number analyzed (Participants) | 50 | 50 | 29
scores on a scale
  Baseline | 3.8 (0.7) | 4.0 (0.6) | 4.1 (0.5)
  6 months: number analyzed (Participants) | 44 | 47 | 0
  6 months | 4.0 (0.7) | 3.9 (0.7) |
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48 | 27
  End of Study at 12 Months Post-Randomization | 3.9 (0.7) | 3.9 (0.6) | 4.1 (0.5)

4. Secondary Outcome: Health-Related Quality of Life (Type 1 Diabetes and Life)
Description: The Type 1 Diabetes and Life (T1DAL) measure assesses diabetes-specific health-related quality of life. Participants will complete the T1DAL version for their age (Adolescent: 12-17, 23 items; Young Adult: 18-25, 27 items; Adult-1: 26-45, 27 items), which asks respondents to rate the degree to which each item is true about their everyday quality of life with diabetes. Items responses range from 1 (not at all true) to 5 (very true). Total scores are calculated by reverse-scoring items as indicated in the measure development paper instructions, then calculating a mean score and multiplying by 25 to convert the scores to a 100 point scale. The lowest possible total score is 0 and the highest possible total score is 100. Higher total scores = better T1D-specific health-related quality of life overall.
  Collected for young adult participants in both arms (baseline and 12 mo) and Peer Mentors (pre- and post-involvement in study).
Time Frame: Baseline and End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care | Peer Mentors
Number analyzed (Participants) | 50 | 50 | 29
scores on a scale
  Baseline | 65.5 (15.8) | 66.7 (15.4) | 65.6 (12.5)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 47 | 27
  End of Study at 12 Months Post-Randomization | 68.4 (16.0) | 63.0 (14.6) | 61.6 (14.5)

5. Secondary Outcome: Diabetes Strengths (Diabetes Strengths and Resilience Measure)
Description: The Diabetes Strengths and Resilience (DSTAR) measure assesses participants' self-perceptions about what they do well with diabetes (known as diabetes strengths). Participants will complete the Young Adult version of the DSTAR, which asks respondents to rate how often the items represent their experiences/perspectives about their diabetes strengths. Items responses range from 0 (never) to 4 (almost always). A total score is calculated by summing the 16 item responses. Lowest possible total score = 0, highest possible total score = 64. Higher total scores = more diabetes strengths.
  Collected for young adult participants in both arms, not Peer Mentors.
Time Frame: Baseline, 6-Month Post-Randomization, & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care
Number analyzed (Participants) | 50 | 50
scores on a scale
  Baseline | 50.4 (10.1) | 50.0 (9.3)
  6 months: number analyzed (Participants) | 44 | 47
  6 months | 52.1 (9.2) | 49.7 (9.4)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  End of Study at 12 Months Post-Randomization | 52.8 (8.6) | 50.1 (10.4)

6. Secondary Outcome: Social Support (Brief 2-Way Social Support Scale)
Description: The Brief 2-Way Social Support Scale (Brief-2SSS) is a 12-item measure that assesses experiences of giving and receiving social support. There are 4 scales: giving emotional support, giving instrumental support, receiving emotional support, receiving instrumental support. Items responses range 0 (not at all) to 5 (always). Higher scores = higher perceived support.
  Young adults complete all subscales at baseline and 12 months, and only the 2 "Receiving" subscales at 6 months. Peer Mentors completed all 4 subscales. A Total score (combined) is calculated by summing all items, Range 0-60.
  Collected for young adult participants in both arms (baseline & 12 mos) and Peer Mentors (pre- and post-involvement in study).
Time Frame: Baseline & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care | Peer Mentors
Number analyzed (Participants) | 50 | 50 | 29
scores on a scale
  Baseline | 50.2 (7.0) | 46.5 (9.0) | 52.1 (4.5)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48 | 27
  End of Study at 12 Months Post-Randomization | 50.3 (7.9) | 47.1 (10.0) | 52.7 (5.4)

7. Secondary Outcome: Diabetes Distress (Diabetes Distress Scale for Adults With T1D)
Description: The Diabetes Distress Scale for Adults with T1D (DDS-T1D) is a 28-item self-report scale that measures participants' experiences with distress related to living with diabetes. It assesses seven dimensions of distress: powerlessness, management distress, hypoglycemia distress, negative social perceptions, eating distress, physician distress, and friends/family distress. Items responses range from 1 (not a problem) to 6 (a very serious problem). The total DDS-T1 score is calculated by averaging the items . Min possible total score = 1, Max = 6. Higher scores = more diabetes distress; average score <2.0 = little/no distress, 2.0-2.9 = moderate distress, 3.0 or higher = high distress.
  Collected for young adult participants in both arms (baseline, 6 mo, 12 mo) and Peer Mentors (pre- and post-involvement in study).
Time Frame: Baseline, 6-Month Post-Randomization, & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
  1 missing value at baseline due to scoring rules, unable to calculate a total score due to missing data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care | Peer Mentors
Number analyzed (Participants) | 49 | 50 | 29
scores on a scale
  Baseline | 2.3 (1.0) | 2.0 (0.7) | 1.8 (0.6)
  6 months: number analyzed (Participants) | 44 | 47 | 0
  6 months | 1.8 (0.8) | 2.0 (0.7) |
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48 | 27
  End of Study at 12 Months Post-Randomization | 1.7 (0.7) | 2.0 (0.8) | 1.8 (0.6)

8. Secondary Outcome: Depressive Symptoms (PROMIS Short Form Depression 4a)
Description: The PROMIS Short Form Depression 4a consists of 4 items that are pulled from the PROMIS Depression Item Bank v1.0. These items assess how often the individual has been bothered by depression-related symptoms, including negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), and decreased positive affect and engagement (loss of interest, meaning, and purpose), over the last 7 days. Items responses range from 1 (never) to 5 (always). A total score is calculated by summing the items, ranging from 4-20. Higher scores = more depressive symptoms.
  Collected for young adult participants in both arms, not Peer Mentors.
Time Frame: Baseline, 6-Month Post-Randomization, & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care
Number analyzed (Participants) | 50 | 50
scores on a scale
  Baseline | 7.3 (4.2) | 7.2 (3.6)
  6 months: number analyzed (Participants) | 44 | 47
  6 months | 6.0 (3.1) | 8.0 (4.1)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  End of Study at 12 Months Post-Randomization | 7.1 (4.0) | 7.5 (4.2)

9. Secondary Outcome: Emotional Support (PROMIS Short Form Emotional Support 4a)
Description: The PROMIS Short Form Emotional Support 4a assesses perceived feelings of being cared for and valued as a person and having supportive relationships. Participants respond to 4 items on a scale from 1(Never) to 5 (Always) . A total score is calculated by summing the items. The possible range is 4-20. Higher scores = more perceived emotional support.
  Collected for young adult participants in both arms, not Peer Mentors.
Time Frame: Baseline, 6-Month Post-Randomization, & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care
Number analyzed (Participants) | 50 | 50
scores on a scale
  Baseline | 16.7 (4.3) | 16.8 (3.8)
  6 months: number analyzed (Participants) | 44 | 47
  6 months | 17.5 (3.1) | 16.8 (3.7)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  End of Study at 12 Months Post-Randomization | 17.6 (2.7) | 16.4 (3.8)

10. Secondary Outcome: Informational Support (PROMIS Short Form Informational Support 4a)
Description: The PROMIS Short Form Informational Support 4a assesses perceptions about the information or resources others provide to them (adequacy, availability, helpfulness). Participants respond to 4 items on a scale from 1(Never) to 5 (Always). A total score is calculated by summing the items. The possible range is 4-20. Higher scores = more perceived informational support.
  Collected for young adult participants in both arms, not Peer Mentors.
Time Frame: Baseline, 6-Month Post-Randomization, & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care
Number analyzed (Participants) | 50 | 50
scores on a scale
  Baseline | 16.2 (4.0) | 15.9 (3.9)
  6 months: number analyzed (Participants) | 44 | 47
  6 months | 17.2 (2.9) | 16.5 (3.4)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  End of Study at 12 Months Post-Randomization | 17.0 (3.5) | 16.3 (4.0)

11. Secondary Outcome: Social Isolation (PROMIS Short Form Social Isolation Item)
Description: The PROMIS Short Form Social Isolation item is a single-item measure from the PROMIS item bank that assesses participants' feelings of being isolated from other people. There is no time frame for responding to this measure. Participants respond to 1 item on a scale from 1 (Never) to 5 (Always), which is equivalent to the total score (higher = more perceived isolation).
  Collected for young adult participants in both arms (baseline, 6, & 12 mos), not Peer Mentors.
Time Frame: Baseline, 6-Month Post-Randomization, & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care
Number analyzed (Participants) | 50 | 50
scores on a scale
  Baseline | 2.6 (1.3) | 2.5 (1.1)
  6 months: number analyzed (Participants) | 44 | 47
  6 months | 2.2 (1.1) | 2.8 (1.3)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  End of Study at 12 Months Post-Randomization | 2.5 (1.1) | 2.5 (1.3)

12. Secondary Outcome: Transition Readiness (Readiness Assessment of Emerging Adults With Type 1 Diabetes Diagnosed in Youth)
Description: The Readiness Assessment of Emerging Adults With Type 1 Diabetes Diagnosed in Youth (READDY) is a 46-item self-report scale that measures participants' preparation for the transition to adult diabetes care, including: knowledge of diabetes, navigation of diabetes care, management skills and behaviors, and insulin pump skills if applicable. Only 18 items from the 3 subscales [Knowledge (4 items - baseline and 12 mos only), Navigation (13 items, baseline, 6 and 12 mos), Health Behaviors (1 item, baseline and 12 mo only)] will be administered for this study. Items responses range from 0 (haven't thought about it) to 5 (yes, I can do this). For each subscale, a subscale score is calculated by averaging the items. Possible score range for each subscale = 1-5. Higher scores = higher readiness in each domain.
  Collected for young adult participants in both arms (baseline, 6, & 12 mos), not Peer Mentors.
Time Frame: Baseline, 6-Month Post-Randomization, & End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care
Number analyzed (Participants) | 50 | 50
scores on a scale
  Knowledge Scale - Baseline | 3.9 (1.0) | 3.9 (1.1)
  Knowledge Scale - 6 months: number analyzed (Participants) | 44 | 47
  Knowledge Scale - 6 months | 4.3 (0.8) | 4.0 (1.2)
  Knowledge Scale - End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  Knowledge Scale - End of Study at 12 Months Post-Randomization | 4.4 (0.8) | 4.0 (1.1)
  Navigation Scale - Baseline | 4.3 (0.6) | 4.3 (0.8)
  Navigation Scale - 6 months: number analyzed (Participants) | 44 | 47
  Navigation Scale - 6 months | 4.5 (0.6) | 4.3 (0.8)
  Navigation Scale - End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  Navigation Scale - End of Study at 12 Months Post-Randomization | 4.7 (0.5) | 4.4 (0.7)
  Health Behaviors Scale - Baseline | 4.8 (0.6) | 4.7 (1.0)
  Health Behaviors Scale - 6 months: number analyzed (Participants) | 44 | 47
  Health Behaviors Scale - 6 months | 4.8 (0.4) | 4.7 (0.9)
  Health Behaviors Scale - End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  Health Behaviors Scale - End of Study at 12 Months Post-Randomization | 4.9 (0.4) | 4.6 (1.1)

13. Secondary Outcome: General Quality of Life (Satisfaction With Life Scale)
Description: The Satisfaction with Life Scale (SWLS) is a 5-item self-report scale that measures participants' perceptions about their life overall. Items responses range from 1 (strongly disagree) to 7 (strongly agree). A total score is calculated by summing the items. Possible score range = 5-35. Higher = greater overall satisfaction with life.
  Collected for young adult participants in both arms (baseline and 12 mo), not Peer Mentors.
Time Frame: Baseline and End of Study at 12 Months Post-Randomization
Population: Differences between total analyzed and analyzed at follow-ups is due to participant attrition
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DiaBetter Together Intervention | Usual Care
Number analyzed (Participants) | 50 | 50
scores on a scale
  Baseline | 23.1 (8.1) | 24.0 (6.7)
  End of Study at 12 Months Post-Randomization: number analyzed (Participants) | 44 | 48
  End of Study at 12 Months Post-Randomization | 24.0 (8.5) | 22. (6.8)

ADVERSE EVENTS:
Time Frame: Consent through completion of final study follow-up (12 months plus up to 3 month data collection window)
Groups:
- DiaBetter Together Intervention: Young Adult participants with type 1 diabetes (ages 17-25) who are approaching transfer from pediatric to adult care will be randomized to either the DiaBetter Together Intervention group or the Usual Care group. After randomization to the intervention group, young adults will be assigned a Peer Mentor. Following an intervention manual, the Peer Mentor will teach behavioral strategies and offer support to the young adult. In both conditions, participation in this study will not impact participants' ability to contact the pediatric care team or other medical services to receive care.
  DiaBetter Together: Following a manual, the Peer Mentor will teach behavioral strategies and offer support to the young adult, including (a) teaching and modeling strengths-based skills for goal-setting, problem-solving, stress management; (b) guiding participants in obtaining support from their social support network (e.g., family, friends); (c) developing a plan for accountability around diabetes management and follow-up in adult care; (d) sharing transition experiences and strategies for successfully navigating the adult healthcare system; (e) discussing how to prioritize diabetes self-care; and (f) assisting them in accessing diabetes-related resources (e.g., local diabetes groups, apps, social media). Contact will be in-person, by phone, email, text message, and/or video, approximately weekly for first 3 mos, approximately biweekly for next 3 mos, and approximately monthly for last 6 mos
Arm/Group | DiaBetter Together Intervention | Peer Mentors | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/29 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/29 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/29 | 0/50

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, participant accrual was delayed and resulted in a smaller randomized sample size (n=100) than anticipated (n=150) Some measures listed as Outcome measures section (e.g., sleep, COVID-19 experiences , stressful events) were not primary or secondary outcomes of the trial, but rather descriptive or exploratory measures, and thus were not included in the Outcome Measures results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT04247620/Prot_SAP_000.pdf